CLINICAL TRIAL: NCT06424548
Title: A Randomized, Open-label, Investigator-initiated, Pilot Clinical Trial Comparing the Improvement for Ankle Brachial Index and Safety of Sarpogrelate and Clopidogrel in Stroke Patients Accompanying Lower Extremity Vascular Atherosclerosis With Decrease of Ankle Brachial Index and Intermittent Claudication.
Brief Title: Comparison of the Improvement and Safety of the Ankle Brachial Arterial Pressure Index of Sarpogrelate and Clopidogrel in Stroke Patients With Decreased Ankle Brachial Arterial Pressure Index and Intermittent Claudication of Lower Limb Vascular Atherosclerosis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ewha Womans University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Tae-Jin Song, MD, PhD, Principal Investigator, Ewha Womans University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEUMC 2023-10-009
Record Dates: First submitted 2024-04-15; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Atherosclerosis
MeSH Terms: conditions — Stroke; Atherosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of Sarpogrelate (Experimental): The intervention group will receive aspirin 100mg plus sarpogrelate 100mg
  Interventions: Drug: Administration of Sarpogrelate
- Traditional administration of Clopidogrel (Other): The control group will receive aspirin 100mg plus clopidogrel 75mg
  Interventions: Drug: Traditional administration of Clopidogrel

INTERVENTIONS:
Drug: Administration of Sarpogrelate — Aspirin 100mg plus Sarpogrelate 100mg
  Arms: Administration of Sarpogrelate
Drug: Traditional administration of Clopidogrel — Aspirin 100mg plus Clopidogrel 75mg
  Arms: Traditional administration of Clopidogrel

SUMMARY:
The clinical trial aims to confirm the improvement effect of the ankle brachial index and the safety of sarpogrelate administration compared to clopidogrel in stroke patients with decreased ankle brachial arterial pressure index and intermittent claudication of lower limb vascular atherosclerosis. Subjects are assigned to one of the two combinations through random allocation.

Intervention group: Aspirin 100mg + sarpogrelate 300mg dosing group, Control group: Aspirin 100mg + clopidogrel 75mg dosing group. This clinical trial is a prospective open study and will be conducted in compliance with the usual diagnosis and treatment process, and in particular, all trial subjects will be tested and treated appropriately in accordance with the standard treatment guidelines for ischemic stroke during the clinical trial period.

DETAILED DESCRIPTION:
A total of 100 subjects are recruited and divided into a intervention group and a control group through randomization.

In this clinical trial, the intervention group and the control group are assigned 1:1.

The researcher allocates 1:1 to the intervention group or control group through a two-way random number table on the assignment date in the order of the subjects who are satisfied with the Inclusion and exclusion criteria and agreed to the study.

This study is a prospective open randomized clinical trial that can confirm which group the subjects themselves were assigned to. After randomization, the drug is prescribed and the outcome variable is checked at 12 months.

During the course of the clinical trial, the examiner and researchers carefully observe the presence or absence of adverse events during the follow-up period after randomization, and closely observe outcome variables, including neurological changes.

Visit after 6 months and 12 months during the clinical trial period to confirm the effectiveness and safety. When an event corresponding to the outcome variable occurs, the researcher first plans to implement appropriate medical measures in this regard.

Both groups will be conducted in compliance with the usual diagnosis and treatment process, and in particular, all subjects will be tested and treated appropriately according to the standard treatment guidelines for ischemic stroke during the clinical trial period.

The purpose of this study is to determine whether there is a difference in the improvement and safety of the ankle-brachial arterial pressure index of aspirin+sarpogrelate and aspirin+clopidogrel in stroke patients with decreased ankle-brachial arterial pressure index and intermittent claudication.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 or over.
2. Neurologically stable patients after 7 days and within 6 months of diagnosis of ischemic stroke.
3. Patients with ankle-brachial index (ABI) <0.9 performed within 6 months of screening, with lower limb vascular stenosis and intermittent claudication.
4. A person who voluntarily agrees to participate in this clinical trial in writing.

Exclusion Criteria:

1. Patients who are unable or contraindicated to administer antithrombotic drugs.
2. Patients with less than 80,000 platelets, less than 8.0 hemoglobin, liver levels and total bilirubin levels three times normal according to laboratory standards, according to blood tests conducted within one month.
3. Patients identified as undergoing renal replacement therapy such as dialysis due to acute or terminal nephropathy during screening.
4. Patients diagnosed with or treated for cancer within 6 months of screening, or identified as having recurrent or metastatic cancer.
5. Patients confirmed to be on medication for liver diseases such as liver cirrhosis during screening.
6. A pregnant and lactating women.
7. Patients with a history of hemorrhagic tendency, conventional cerebral hemorrhage, and gastrointestinal hemorrhage.
8. Patients who need oral anticoagulant therapy instead of antiplatelet drugs for screening.
9. Patients who are at least 3 in the Rutherford category and need lower-limb vascular procedure/surgery within 6 months, as judged by the doctor.
10. A patient with a loss of consciousness/cognition.
11. Any person who determines that the tester is not suitable for participating in the clinical trial for other reasons.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-16 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Ankle brachial index | Baseline, 12months
  The value of the ankle brachial index evaluated 12 months after the first dose of the clinical trial drug. Ankle brachial index : normal range > 0.9, abnormal range < 0.9

SECONDARY OUTCOMES:
Ankle brachial index | Baseline, 6months
  The value of the ankle brachial index evaluated 6 months after the first dose of the clinical trial drug. Ankle brachial index : normal range > 0.9, abnormal range < 0.9
Brachial ankle pulse wave velocity | Baseline, 6months, 12months
  The value of Brachial ankle pulse wave velocity evaluated 6 months and 12months after the first dose of the clinical trial drug. Brachial ankle pulse wave velocity : normal range 1000~1500 cm/sec, abnormal range > 1600 cm/sec
Major cardio-cerebrovascular events | Baseline, 6months, 12months
  Major cardio-cerebrovascular events that occurred within 6 months and 12 months after the first medication related to the clinical trial. (Stroke, myocardial infarction, non-stable angina, lower limb vascular intervention, surgery, death)
Lower limb angioplasty or re-operation | Baseline, 6months, 12months
  Whether or not to perform lower limb angioplasty or re-operation, evaluated 6 months and 12 months after the first dose of the clinical trial drug.
Change of Rutherford category ratio | Baseline, 6months, 12months
  Change of Rutherford category ratio, a symptom scale related to vascular stenosis of the lower extremities, evaluated 6 months and 12 months after the first dose of the clinical trial drug. (Grade 0-Asymptomatic, Grade 1-Mild claudication, Grade 2-Moderate claudication, Grade 3-Severe claudication, Grade 4-Ischemic rest pain, Grade 5-Minor tissue loss-nonhealing ulcer, focal gangrene with diffuse pedal ischemia, Grade 6-Major tissue loss-extending above transmetatarsal level, functional foot no longer salvageable)
Modified Rankin scale | Baseline, 6months, 12months
  Modified Rankin scale evaluated 6 months and 12 months after the first dose of the clinical trial drug. (0-No symptoms at all, 1-No significant disability despite symptoms; able to carry out all usual duties and activities, 2-Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance, 3-Moderate disability; requiring some help, but able to walk without assistance, 4-Moderate to severe disability; unable to walk without assistance, and unable to attend to own bodily needs without assistance, 5-Severe disability; bedridden, incontinent and requiring constant nursing care and attention, 6-Death)
National Institutes of Health Stroke Scale | Baseline, 6months, 12months
  Changes in NIHSS evaluated at 6 months and 12 months after the first dose of the clinical trial drug. National Institutes of Health Stroke Scale score of 0 (lowest point) means normal, and a score of 42 (high point) means severe dysfunction caused by stroke, so the higher the score, the more severe the stroke.
Coronary angioplasty | Baseline, 6months, 12months
  Confirmation that coronary angioplasty was performed at 6 months and 12 months after the first dose of the drug in the clinical trial.
Cerebrovascular angioplasty | Baseline, 6months, 12months
  Confirmation that cerebrovascular angioplasty was performed at 6 months and 12 months after the first dose of the drug in the clinical trial.

IPD SHARING:
Plan to Share IPD: No